CLINICAL TRIAL: NCT04957303
Title: Machine Learning-assisted Analysis of Microcirculation Patterns and Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202003094RINA
Record Dates: First submitted 2021-06-23; First posted 2021-07-12 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Sublingual Microcirculation Pattern and Parameter Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sublingual microcirculation video recording — The sublingual microcirculation videos were recorded by video microscope

SUMMARY:
Machine learning has been widely used in clinical medicine in recent years. It can be used for disease classification, disease severity grading, genetic testing, image analysis, adjuvant treatment recommendations, and predicting patient prognosis. Because sublingual microcirculation can be used for guiding shock resuscitation, a real time automated analysis is required for rapid changes of clinical condition. This study aims to use machine learning to analyze the parameters and patterns of sublingual microcirculation.

DETAILED DESCRIPTION:
The sublingual microcirculation videos are extracted from the 11 clinical trials conducting in the National Taiwan University Hospital.

In the first stage, the microcirculation videos and the related information are included in a de-identified manner. Each microcirculation video in the database will have a unique code. The video-related data will include the patient's height, weight, blood pressure, heartbeats, health status, major diseases, laboratory examination values, video quality description, automated vascular analysis (AVA) 3 software analysis results including total vessel density (TVD), perfused vessel density (PVD), proportion of perfused vessels (PPV), microvascular flow index (MFI), and heterogeneity index (HI). The length of each micro-cycle video is 4-6 seconds, and there are 25 frames per second. Take a picture as a representative image, each video can correspond to 4 images, and each micro-circulation image will also be marked with its image quality. Machine learning model will be trained for distinguishing the quality of videos and images. Only good-quality videos and images will be used for further analysis.

In the second stage, 80% of the microcirculation videos and images will be used for training and validation to find the best model, and then the remaining 20% of microcirculation videos and images will be used to test the model performance. The first training purpose is to automatically distinguish the size of blood vessels, calculate TVD, and draw a histogram of the number of microvessels of different diameters. The second training purpose is to measure the blood flow velocity in each small vessel and calculate PVD, MFI, and HI values.

ELIGIBILITY:
Inclusion Criteria:

* Microcirculation videos and images from previous clinical trials in the National Taiwan University Hospital with signed informed consent and agreement of further analysis

Exclusion Criteria:

* Microcirculation videos and images from previous clinical trials in the National Taiwan University Hospital with signed informed consent but disagreement of further analysis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers Critically ill patients Surgical patients Patients with dialysis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Perfused vessel density | 6 seconds
  Training machine learning models to view the videos of patients' sublingual microcirculation images and calculate the perfused vessel density. The videos of patients' sublingual microcirculation images are obtained and recorded by the video microscopes.

SECONDARY OUTCOMES:
Patterns of microcirculation | 6 seconds
  Training machine learning models to view the videos of patients' microcirculation images and distinguish the patterns of microcirculation images and videos among healthy volunteers and patients with specific diseases or clinical conditions (eg. dialysis, postoperative, or septic shock.) The videos of patients' sublingual microcirculation images are obtained and recorded by the video microscopes.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No